CLINICAL TRIAL: NCT06131424
Title: Multicentre NIS Retrospective Study to Know the Prevalence of HER2- Low,Clinical Characteristics,Treatment Patterns,Associated Outcome in Patient With HER2-negative in Metastatic Breast Cancer Who Progressed on Systemic Anticancer Therapy
Brief Title: NIS Study Determining Prevalence of HER2-low in Metastatic Breast Cancer Patients
Acronym: iRetroBC
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9673R00037
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: HER2-negative
Keywords: HER2 Low, Metastatic breast cancer; HR:Hormone Receptor, IHC:mmunohistochemistry; ISH: in situ hybridization; Anticancer therapy; Prognostic and Predictive Biomarker; Formalin-fixed, paraffin-embedded (FFPE); endocrine therapy(ET); Subsets
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This noninterventional, multicenter,retrospective study has been proposed to estimate the prevalence, clinicopathological characteristics,treatment patterns and clinical outcomes of human epidermal growth factor receptor 2 -(HER2)low locally-advanced or metastatic breast cancer(mBC) by accurate rescoring of archived IHC-stained formalin-fixed paraffin-embedded (FFPE) slides for HER2 in patients previously identified as HER2-negative from emerging markets of international regions (non-US and non-European region) with largely unknown prevalence estimates of HER2 low mBCs. Patients with a confirmed diagnosis of HER2-negative, locally-advanced or mBC regardless of Hormone receptor (HR)status between 01 January 2019 and 31 December 2022 who progressed on any systematic anticancer therapy (eg, ET, chemotherapy, CDK4/6 inhibitor, targeted therapies other than anti-HER2, or immunotherapy) in advanced disease with availability of atleast 12 months of follow-up data (from the index date) in the medical records at the participating site, unless patient died within the first 12 months of diagnosis of locally-advanced or mBC will be enrolled in the study. The HR positive patients will be considered eligible for the study if they have received ET as adjuvant therapy in the early BC setting and progressed within 24 months. This scenario will be considered as progression on systematic treatment in the advanced or metastatic setting.

DETAILED DESCRIPTION:
Multicenter, noninterventional, retrospective study, aimed to determine the prevalence of HER2-low and HER2>0<1+ by rescoring of archived IHC-stained FFPE slides for HER2 in patients previously identified as having HER2-negative locally-advanced or mBC who progressed on any systemic anticancer therapy.The study will also describe the baseline sociodemographic and clinicopathological characteristics, treatment patterns, clinical outcomes and concordance between historical IHC status and rescored IHC status of archived IHC-stained FFPE slides. The study will not have any study-specific patient visits, procedures, or a longitudinal follow-up. All available data will be extracted from patients' medical records. The study will consist of 2 components: rescoring of archived IHC-stained FFPE slides and secondary data collection from patients' medical records. Human epidermal growth factor receptor 2 IHC historical scores, HER2 rescoring results of archived IHC-stained FFPE slides by qualified laboratory (local and/or independent central laboratory), other biomarker testing results based on historical testing and/or testing of archived tissue samples when available. The data on different types of treatment received by the patients and sociodemographics and clinicopathological characteristics will be extracted from patients' medical records from the date of diagnosis of HER2-negative BC up to the date of data extraction.

The patients identified for the current study will be a convenience sample of all patients in the relevant electronic health record/electronic medical record databases and biobanks who meet the inclusion and exclusion criteria; no a priori power analysis will be conducted. The study aims to capture approximately minimal 150 to 200 HER2-negative mBC patients per participating country/cluster, in order to generate data on 2100 to 2700 patients overall, with the aim to identify approximately 1050 HER2-low patients (at least 600 patients in Asia cohort and 450 patients in Latin America [LATAM] cohort) for analysis, subject to revision based on preliminary data analysis. Clinical outcomes will be assessed as per the HER2 subsets identified after rescoring (HER2 low-IHC1+ or IHC2+/ISH-, HER2 IHC>0<1+, HER2 null, and HER2 zero-HER2 IHC>0<1+ and HER2 null). The study will be conducted in 8 Asian countries including Hong Kong, India, Indonesia, Malaysia, Philippines, Thailand, Singapore, and Vietnam and 6 Latin American (LATAM) countries including Argentina, Brazil, Chile, Dominican Republic, Mexico, and Panamá. Regions and countries may be added based on feasibility assessment as per AstraZeneca's standard operating procedures. A total of approximately 2100 to 2700 patients with a confirmed diagnosis of HER2-negative, locally-advanced or mBC regardless of HR status between 01 January 2019 and 31 December 2022 with the availability of medical records of at least 12 months of follow-up data (from the index date), and deemed eligible as per the study eligibility criteria will be enrolled in the study at approximately 28-58 study sites. The study protocol and informed consent form (ICF) will be approved by local Institutional Review Boards (IRBs)/(Institutional) Ethics Committees (IECs) before the commencement of recruitment.

ELIGIBILITY:
Inclusion Criteria:1. Men or women, ≥18 years of age 2. Provision of informed consent by the patient or next of kin/legal representative (for deceased patients at study entry, unless a waiver was granted) according to local regulations 3. Must have a histological or cytological confirmed previous diagnosis as HER2-negative (IHC zero, 1+, 2+/ISH-) locally-advanced or mBC between 01 January 2019 and 31 December 2022, regardless of HR status 4. Must have progressed on any systemic anticancer therapy (eg, ET, chemotherapy, CDK4/6 inhibitor, targeted therapies other than anti-HER2, or immunotherapy) in the metastatic setting with the availability of at least 12 months of follow-up data (from the index date) in the medical records at the participating site, unless patient died within the first 12 months of diagnosis a) The HR positive patients will be considered eligible for the study if they have received ET as adjuvant therapy in the early BC setting and progressed within 24 months, this scenario will be considered as progression on systematic treatment in the advanced or metastatic setting 5. Must have historical IHC-stained FFPE tissue from locally-advanced or mBC slides for HER2 in an acceptable quality to allow for accurate rescoring of HER2 expression - Exclusion Criteria:1. Have a history of other malignancies, other than basal cell carcinoma of the skin and squamous cell carcinoma of the skin until 3 years prior to diagnosis of locally-advanced or mBC 2. Patients with historical HER2 status of IHC 2+/ISH+ or 3+, or HER2 amplified

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients from sites will be selected in a consecutive manner ie, patients with dates closest to but on or after 01 January 2019 will be selected first.
Sampling Method: Probability Sample
Enrollment: 1151 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with IHC 1+ or IHC 2+/ISH- HER2 expression. | 6 months from the Last subject In
  1. Proportion of patients with IHC 1+ or IHC 2+/ISH- HER2 expression among previously identified HER2-negative locally-advanced or mBC patients based on rescoring of archived IHC-stained FFPE slides.
Proportion of patients with HER2 ultra-low (IHC 0 (pattern 0+) with membrane staining ie, incomplete and faint/barely perceptible in ≤10% tumor cells) HER2 expression and IHC null (IHC 0 ie, absent membrane staining), | 6 months from the Last subject In
  Proportion of patients with HER2 ultra-low (IHC 0 (pattern 0+) with membrane staining ie, incomplete and faint/barely perceptible in ≤10% tumor cells) HER2 expression and IHC null (IHC 0 ie, absent membrane staining), expanded biomarker association with HER2-low patient characteristics, change in HER2 and HR expressions between diagnosis and treatment, concordance of HER2 IHC scores between manual rescoring and digital scoring.

SECONDARY OUTCOMES:
Sociodemographic (age, gender, smoking status, country, ethnicity, site type [community hospital, academic hospital, biobank, research institute], family history of BC) and clinical pathological characteristics | 6 months from the Last subject In
  Menopausal status
  * Age at initial diagnosis of BC
  * Eastern Cooperative Oncology Group (ECOG) performance status (0 = fully active to 4 = completely disabled) at index date
  * Tumor, nodes, metastases (TNM) staging at initial diagnosis of BC and locally-advanced or mBC stage
  * Tumor grade at first diagnosis, and at index date (if available)
  * HR status (ER/PR - positive/negative)
  * BRCA mutation status
  * Histological type (ductal, lobular, mixed, other)
  * Comorbidities (diabetes mellitus, hypertension, cardiovascular disease, osteoporosis)
  * Treatment for early-stage BC with duration (if available)
  * Locoregional treatment received (yes/no) after index date • Diagnostic tests/investigations (radiological, laboratory)
  * Oncotype or MammaPrint status/results (if available) • Endocrine refractory/sensitive status (if available) • Date of diagnosis and duration of each LOT in locally-advanced or mBC setting
Proportions of patients in the overall study population and each study subset receiving the following treatments for early-stage BC (if available), locally-advanced or mBC | 6 months from the Last subject In
  Anti-HER2 targeted therapy ([Antibody: trastuzumab, pertuzumab], [ADC: trastuzumab emtansine, T-DXd], [tyrosine kinase inhibitor: lapatinib, neratinib, and tucatinib])
  * Standard chemotherapy
  * Hormonal/endocrine therapies (aromatase inhibitor, alpelisib, ethinyl estradiol, fluoxymesterone, megestrol acetate, fulvestrant [selective ER degrader, SERD], tamoxifen)
  * Immunotherapy
  * Targeted therapy (CDK4/6 inhibitor, everolimus, AKT inhibitor)
  * Other
Clinical outcomes | 6 months from the Last subject In
  Following outcomes for locally-advanced or mBC in the overall study population and HER-2 subsets identified after rescoring (HER2 low-IHC1+ or IHC2+/ISH-, HER2 IHC>0<1+; HER2 null, and HER2 zero-HER2 IHC>0<1+ and HER2 null). (a) Median OS Following outcomes will also be assessed by each LOT (b) Median TFST and Median TTD (c) Median rwPFS (d) rwORR
Concordance between rescoring IHC status as HER2-low by central laboratory and/or local laboratory | 6 months fromthe last subject In
  Historical scoring and local laboratory rescoring of HER2 IHC status

OTHER OUTCOMES:
Summary of the following biomarkers using available historical next generation sequencing (NGS) or IHC results | 6 months from the Last subject In
  ER, PR status (positive or negative) and % of cells with Nuclear positivity (if available) and average intensity of staining (if available) • Ki-67 in % nuclei (if available) • PD-L1 IHC and methodology (if available) • PIK3CA gene mutations • ESR1 gene mutations • BRCA1 and BRCA2 gene mutations • PALB2 gene mutations • AKT1 gene mutations • ATM gene mutations • PTEN gene mutations • Other

CONTACTS AND LOCATIONS:
Locations (23):
- Research Site, Rosario, Argentina
- Research Site, São Paulo, Brazil
- Research Site, Santo Domingo, Dominican Republic
- Research Site, Hong Kong, Hong Kong
- India (8):
  - Research Site, Bengaluru, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Mumbai, Maharashtra
  - Research Site, Bhubaneshwar, Odisha
  - Research Site, Mohali, Punjab
  - Research Site, Hyderabad, Telangana
  - Research Site, Varanasi, Uttar Pradesh
  - Research Site, Delhi
- Research Site, Jakarta, Indonesia
- Malaysia (2):
  - Research Site, Kaula Lumpur
  - Research Site, Subang Jaya
- Research Site, Mexico City, Mexico
- Research Site, Panama City, Panama
- Research Site, Quezon City, Philippines
- Research Site, Singapore, Singapore
- Research Site, Bangkok, Thailand
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home